CLINICAL TRIAL: NCT03916614
Title: Relief of Symptoms of Post-traumatic Stress for Victims of Gun Violence:
Brief Title: Relief of Symptoms of Post-traumatic Stress for Victims of Gun Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000025580
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: PTSD; Stress, Psychological; Gunshot Wound
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Stress, Psychological; Wounds, Gunshot | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- START treatment (Experimental): Participants randomized into the treatment arm will receive the START intervention as described above alongside usual care from the VPOP staff
  Interventions: Behavioral: Screening Tool for Relief of Trauma (START)
- standard of care (Active Comparator): Those randomized to the control arm will receive the usual screening for PTSD and referral for outpatient services if warranted as well as usual care from VPOP staff.
  Interventions: Behavioral: standard of care

INTERVENTIONS:
Behavioral: Screening Tool for Relief of Trauma (START) — The Screening and Tool for Awareness and Relief of Trauma (START) was developed for patients that come from communities with sustained and persistent trauma. It consists of six screening questions adapted from the validated Primary Care PTSD Screen,[30] with input from focus groups, surveys and in-depth interviews with victims of violence. The full START intervention requires 30-45 minutes of structured conversation at the end of which the participant leaves with a better understanding of trauma symptoms as well as on-the-spot instruction on a set of techniques designed to alleviate the symptoms of PTSD. Based on the results of their screening, the participant will be offered up to four techniques to alleviate their symptoms
  Arms: START treatment
Behavioral: standard of care — Screening for PTSD and referral for outpatient services if warranted as well as usual care from Violence Prevention and Outreach Program (VPOP) staff.
  Arms: standard of care

SUMMARY:
To test the hypothesis that adult individuals who are victims of gun violence will have decreased symptoms of post-traumatic stress after an individual-level intervention with the Screening and Tool for Awareness and Relief of Trauma (START).

DETAILED DESCRIPTION:
In response to the lack of targeted mental health intervention for gunshot wound survivors, the Screening and Tool for Awareness and Relief of Trauma (START) was developed for patients that come from communities with sustained and persistent trauma. It consists of six screening questions adapted from the validated Primary Care PTSD Screen,[30] with input from focus groups, surveys and in-depth interviews with victims of violence and in particular, boys and young men of color. START has been shown to be effective at decreasing symptoms of PTSD in a one-month follow-up, but it has not been piloted on recently injured victims of gun violence specifically nor has it been tested in a randomized control trial design. A better understanding of the utility of this tool and others like it in victims of violent crime for relief of symptoms of post-traumatic stress and prevention of PTSD would contribute to the larger body of literature on PTSD prevention for victims of gun violence while simultaneously addressing a major need in this community.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of gunshot wound presenting to the Emergency room and/or admitted as inpatient that are eligible for the Violence Prevention and Outreach Program (VPOP).

Exclusion Criteria:

* Patients with severe traumatic brain injury
* Children under the age of 18
* Patients otherwise unable to give consent
* Non-English speaking patients
* Victims of sexual assault
* Patients with history of a severe mental illness and/or those already undergoing treatment for a mental illness by a licensed professional.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
PTSD evaluation | baseline
  Post Traumatic Stress Disorder Checklist - Civilian Version (PCL-C)
Change in PTSD evaluation test scores | 12 weeks
  Post Traumatic Stress Disorder Checklist - Civilian Version (PCL-C) A decrease in PCL-C score greater than or equal to 5 points relative to controls.
Change PTSD evaluation test scores | 6 months
  Post Traumatic Stress Disorder Checklist - Civilian Version (PCL-C) A decrease in PCL-C score greater than or equal to 5 points relative to controls.

CONTACTS AND LOCATIONS:
Overall Officials: James Dodington, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

REFERENCES:
- [Derived] O'Neill KM, Schenck C, Vega P, Gawel M, Dodington J. A pilot clinical trial of the Screening and Tool for Awareness and Relief of Trauma for survivors of gun violence. J Trauma Acute Care Surg. 2024 Apr 1;96(4):641-649. doi: 10.1097/TA.0000000000004121. Epub 2023 Aug 21. PMID 37602906